CLINICAL TRIAL: NCT02593292
Title: Program of Research for the Optimization of a Supervised Patient Pathway for Expectant According to Risk in Obstetrics
Acronym: PROSPERO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 69HCL14_0454
Record Dates: First submitted 2015-10-28; First posted 2015-11-02 (Estimated); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Pregnancy
Keywords: Clinical pathway; Electronic Health Records; Maternal Health Services & administration; Patient Access to Records; Patient Satisfaction; Prenatal Care/methods
MeSH Terms: conditions — Patient Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PROSPERO group (intervention group) (Active Comparator)
  Interventions: Behavioral: PROSPERO
- control group (Placebo Comparator)
  Interventions: Other: control

INTERVENTIONS:
Behavioral: PROSPERO — The intervention is carried out in 3 steps:
  1. At the start of the pregnancy: a number of process steps are defined for a patient's pathway adapted to medical, obstetric and social risk factors.
  2. During pregnancy: city based doctors and midwives work together with their hospital peers enabling patients to participate through the reporting via a medical information system
  3. The entrance in the delivery room: patients are classified as low or high risk for greater vigilance from midwives.
  Arms: PROSPERO group (intervention group)
Other: control — At the start of the pregnancy, medical, obstetric and social risk factors are checked in the same way than the PROSPERO group. An adapted patient pathway was defined by a Clinical Research Assistant but unreachable from patients, midwifes and physicians. The electronic patient care reporting information system will be disabled and midwifes cannot create the classification checklist for low or high risk delivery.
  Arms: control group

SUMMARY:
This French multicentre open-label randomized trial will test the hypothesis that a coordinated health circuit based on obstetric risks, backed up by an electronic patient care reporting information system will optimize the continuum of pregnancy care monitoring. The electronic patient care reporting information system will be shared between patients, private practice physicians/midwifes, hospital physicians/midwifes and supervised by a coordinating midwife.

ELIGIBILITY:
Inclusion Criteria:

* patients over the age of majority,
* enrolled in one of the two maternity hospitals in the study before 12 weeks of amenorrhea (SA) and 6 days (j) of age,
* affiliated to the National Health Insurance Fund of the country within the regional level health insurance
* have an internet access

Exclusion Criteria:

* illiterate patients,
* non-French speakers,
* under the age of majority,
* refusing to participate,
* without internet access,
* followed by one of these maternity wards but delivering else where,
* whose pregnancy ended in a miscarriage early or late (before 21 weeks of amenorrhea (SA) and 6 days (J) over).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1532 (Actual)
Dates: Start 2016-12-05 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-07 (Actual)

PRIMARY OUTCOMES:
Rate of patients'pathway approved as compliant in the intervention group compared to the control group. | at the end of pregnancy
  Compliant patient pathways are those for which all actions (medical visits, examinations, …) recommended during pregnancy, according to the specific risk factors of each patient, will have been made.

SECONDARY OUTCOMES:
rate of severe maternal morbidity and mortality as defined by the EPIdémiologie de la MOrbidité Maternelle Sévère (EPINOMS) project | From 22 completed weeks (154 days) of gestation to seven completed days after birth
rate of perinatal morbidity-mortality as defined by the Organization, Practices Evaluation in perinatal Network | From 22 completed weeks (154 days) of gestation to seven completed days after birth
completeness of all hospital medical records | the end of pregnancy (the date of delivery)
  completeness of hospital medical records compared to electronic patient-reported outcome (ePRO).
health care costs | one week from the date of delivery
  Number of medical visits and hospitalization
health care costs | one week from the date of delivery
  duration of medical visits and hospitalization
patients' satisfaction : Qualitative evaluation by interview | at the end of pregnancy
  Qualitative evaluation of patients' satisfaction and adherence by interview and/or focus groups. Quantitative evaluation of patients' satisfaction and anxiety by the hospital anxiety and depression scale and other validated's patient satisfaction forms
patients' satisfaction : Quantitative evaluation by the hospital anxiety and depression scale | at the end of pregnancy
  Quantitative evaluation of patients' satisfaction and anxiety by the hospital anxiety and depression scale
patients' satisfaction : Qualitative evaluation by interview | within one week from the date of delivery
  Qualitative evaluation of patients' satisfaction and adherence by interview and/or focus groups.
patients' satisfaction : Quantitative evaluation by the hospital anxiety and depression scale | within one week from the date of delivery
  Quantitative evaluation of patients' satisfaction and anxiety by the hospital anxiety and depression scale and other validated's patient satisfaction forms
types of delivery | within one week from the date of delivery
  rate of vaginal delivery, instrumental extraction delivery, Caesarean delivery

CONTACTS AND LOCATIONS:
Overall Officials: René-Charles RUDIGOZ, Pr, Principal Investigator — Hospices Civils de Lyon
Locations (2):
- France (2):
  - Hôpital Femme Mère Enfant, Bron
  - Hospices Civils de Lyon, Lyon

REFERENCES:
- [Background] Gaucher L, Puill C, Baumann S, Hommey S, Touzet S, Rudigoz RC, Cortet M, Huissoud C, Gaucherand P, Dupont C, Mougeot F. The challenge of adopting a collaborative information system for independent healthcare workers in France: a comprehensive study. Sci Rep. 2024 May 19;14(1):11429. doi: 10.1038/s41598-024-62164-2. PMID 38763960
- See also: Related Info — https://hal-hcl.archives-ouvertes.fr/hal-01166092v1